CLINICAL TRIAL: NCT02990520
Title: Prevalence of Malnutrition and/or Sarcopenia at Hospital Admission
Acronym: MASS
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0527
Record Dates: First submitted 2015-09-03; First posted 2016-12-13 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Malnutrition; Sarcopenia
MeSH Terms: conditions — Malnutrition; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the prevalence of malnutrition and/or sarcopenia at admission to the hospital in older adults.

DETAILED DESCRIPTION:
The primary outcome of this study is to determine the prevalence of malnutrition and/or sarcopenia at admission to the hospital in older adults. The secondary outcome is to assess the relationship between malnutrition/sarcopenia status and length of stay, comorbidity load, polypharmacy, and 30-day readmission.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the UTMB ACE unit
* Aged 65 years or older
* Able to consent to participate in study (alert and oriented x3)

Exclusion Criteria:

* Because this study aims to determine prevalence of malnutrition and/or sarcopenia at admission to the hospital, patients will be excluded if study measures are not able to be taken within 72 hours of admission.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized older adults
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of Malnutrition | baseline
  malnutrition measured with questionnaires

SECONDARY OUTCOMES:
Prevalence of sarcopenia | baseline
  Sarcopenia defined using the EWGSOP or IWGS or FNIH criteria

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Principal Investigator — UTMB
Locations (1):
- UTMB Hospitals, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No